CLINICAL TRIAL: NCT06716528
Title: Web-based Application to Test for Long-term Cognitive Deficits in BioCog Patients
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital, Bonn (Other); University Hospital Schleswig-Holstein (Other); Universitätsklinikum Essen (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: BioCog-Web
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Deficits
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Proteomics is emerging as a vital tool in identifying biomarkers of neurodegenerative disease progression and response to therapy. The NUcleic acid Linked Immuno-Sandwich Assay (NULISA)-Seq™ Central Nervous System Disease Panel 120 provides best-in-class sensitivity and robust, multiplexed analysis of 120 neuro-specific and inflammatory proteins from 10 µl of plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Former BioCog patients: Former BioCog patients from the Berlin study center who have undergone baseline cognitive testing and from whom plasma samples are available
- Former BioCog subjects in the non-surgical comparison cohort: Former BioCog subjects in the non-surgical comparison cohort from the Berlin study center who have undergone baseline cognitive testing

SUMMARY:
In the present study, a long-term cognitive follow-up of participants of the BioCog cohort (data collection period 2014 - 2019, Ethical vote No: EA2/092/14) from the Berlin study center is to be will be performed in order to record long-term cognitive sequelae (7 to 10 years after study inclusion). In addition to a medical telephone/video visit, the follow-up includes the collection of cognitive tests via web applications and questionnaires of acceptance and usability in the home environment. The study data are analysed in cooperation with the University of Bonn, University Medical Center Schleswig-Holstein and the University of Essen.

DETAILED DESCRIPTION:
The primary research objective is the exploratory investigation of changes in cognitive test performance as well as cognitive self-care and functionality in former BioCog patients and BioCog subjects in the non-surgical comparison cohort in the long-term follow-up (7 - 10 years) compared to the baseline survey (from the BioCog main study).The primary question is operationalized in several ways:

* according to the International Statistical Classification of Diseases and Related Health Problems(ICD-10) classification system
* according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) classification system
* computer-based, online and independently conducted cognitive testing using Cantab Web based testing from Cambridge Cognition
* Cognitive self-care using Geriatric depression Scale item 10
* Cognitive self-care with Multifactorial Memory Questionnaire
* Cognitive other-care with The Informant Questionnaire on Cognitive Decline in the Elderly questionnaire
* Functionality with Activities of Daily Living (ADLs) & Instrumental Activities of Daily Living (IADLs) questionnaire
* Additionally: Quality of life with 5-level EQ-5D version (EQ-5D-5L)

Evaluation by Mild Cognitive Impairment Algorithm of the University Clinic Bonn (research group Prof. Wagner).

Evaluation by mild/major Neurocognitive Disorder (NCD) algorithm of Charité - University Medicine Berlin (research group Prof. Spies)

ELIGIBILITY:
Patients

Inclusion Criteria:

* Patients of Berliner BioCog cohort with cognitive Testing (CANTAB Research Suite) at Baseline and with plasma samples for baseline that can be contacted.
* Written informed consent for participation in the BioCog-Web study.
* Data and reserve samples from patients in the Berlin BioCog cohort who can no longer be contacted.

Exclusion Criteria:

* None

Subjects

Inclusion Criterion:

-BioCog subjects of the non-operated comparison cohort from Berlin with cognitive testing (CANTAB Research Suite) at baseline who are contactable

Exclusion criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and subjects from the Berlin BioCog cohort.
Sampling Method: Probability Sample
Enrollment: 434 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  The primary object of research is the explorative investigation of the change in cognitive test performance as well as cognitive self-care and functionality in the long-term follow-up (7 - 10 years) compared to the baseline survey (from the main BioCog study). It is measured with CANTAB Research Suite, CANTAB web-based testing and paper pencil tests.

SECONDARY OUTCOMES:
Acceptance | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Acceptance of the CANTAB web-based testing of Cambridge Cognition is measured with a questionnaire.
Usability | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Usability of the CANTAB web-based testing of Cambridge Cognition is measured with a questionnaire.
NUcleic acid Linked Immuno-Sandwich Assay Central Nervous System Disease Multiplex Panel | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Analysis of 120 proteins.
New diagnoses | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Last doctor's letter/last findings (especially in the case of neurological/psychiatric/geriatric connections - e.g. memory consultation) for recording new diagnoses and recording the last outpatient and/or inpatient treatments.
Actual medication | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Current comedication and supplements
Charlson Comorbidity index | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Comorbidity
History of Falls | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  History of falls is measured with the question: Have you had a fall event within the last year?
Depression | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Depression is measured with Geriatric Depression Scale.
Weight history | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Weight history is measured by weight change in the past 3-6 months.
Malnutrition Universal Screening Tool (MUST)-Score | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Add Scores together to calculate overall risk of malnutrition with the Malnutrition screening tool: Score 0 corresponds to low risk; Score 1 corresponds to medium risk; Score 2 or more corresponds to high risk.
Body mass index (BMI) | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  BMI is a calculated measure of a person's body weight (in kilograms) divided by the square of their height (in meters).
Mortality | Participants will be followed for sequelae at 7-10 years after BioCog study inclusion
  Mortality is measured by the number of deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Principal Investigator — Charitè - University Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No